CLINICAL TRIAL: NCT05288452
Title: Food Delivery, Remote Monitoring, and Coaching-Enhanced Education for Optimized Diabetes Management (FREEDOM)
Acronym: FREEDOM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Mississippi Medical Center (Other); Cooper Green Mercy Health Services (Unknown); Pack Health (Industry); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Tapan Shirish Mehta, Professor, Director of Research, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-300008387; 5P50MD017338-03 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-03-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; HIV
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Remote Patient Monitoring

STUDY DESIGN:
Intervention Model Description: We used the multiphase optimization strategy (MOST) as the ideal approach for the proposed study as, with the three proposed intervention components, identifying an optimal intervention through a single randomized controlled trial (RCT) with multiple arms or through multiple RCTs would be methodologically inefficient and resource-intensive. Given this, we rely on the eloquent and rigorous MOST-based optimization design, which leverages factorial experimentation to identify an optimal set of intervention component(s). In a factorial experiment, the goal is not to compare individual experimental conditions (in this case, eight conditions), but to use combinations of conditions to estimate the main and interaction effects of the intervention components. Thus, numerous intervention components can be evaluated simultaneously while utilizing the entire randomized sample.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Arm 1 (Experimental): Digital coaching+ Food delivery+ RPM
  Interventions: Behavioral: Digital Health Coaching; Dietary Supplement: Food Box Delivery; Behavioral: Remote Patient Monitoring (RPM); Behavioral: Diabetes Education Class
- Arm 2 (Active Comparator): Digital coaching
  Interventions: Behavioral: Digital Health Coaching; Behavioral: Diabetes Education Class
- Arm 3 (Active Comparator): Digital coaching+ Food delivery
  Interventions: Behavioral: Digital Health Coaching; Dietary Supplement: Food Box Delivery; Behavioral: Diabetes Education Class
- Arm 4 (Active Comparator): Digital coaching+ RPM
  Interventions: Behavioral: Digital Health Coaching; Behavioral: Remote Patient Monitoring (RPM); Behavioral: Diabetes Education Class
- Arm 5 (Active Comparator): Food delivery+ RPM
  Interventions: Dietary Supplement: Food Box Delivery; Behavioral: Remote Patient Monitoring (RPM); Behavioral: Diabetes Education Class
- Arm 6 (Active Comparator): The participant's will not receive any Intervention
  Interventions: Behavioral: Diabetes Education Class
- Arm 7 (Active Comparator): Food delivery
  Interventions: Dietary Supplement: Food Box Delivery; Behavioral: Diabetes Education Class
- Arm 8 (Active Comparator): RPM
  Interventions: Behavioral: Remote Patient Monitoring (RPM); Behavioral: Diabetes Education Class

INTERVENTIONS:
Behavioral: Digital Health Coaching — The digital health coaching intervention program involves an evidence-based curriculum and one-on-one support to promote positive health behaviors and patient self-management of diabetes.
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Dietary Supplement: Food Box Delivery — The food box intervention component will consist of biweekly food boxes delivered directly to participants over the course of 6 months. The food boxes will contain shelf-stable groceries that adhere to ADA nutritional guidelines for individuals with T2DM.
  Arms: Arm 1; Arm 3; Arm 5; Arm 7
Behavioral: Remote Patient Monitoring (RPM) — The RPM team will instruct the participants to monitor blood glucose levels 3 times daily. Glucose levels will be monitored 8 a.m. to 5 p.m.Monday to Friday. Data summaries will be reviewed bi-monthly with RNs and pharmacists. Participants will be provided with a glucometer, test strips, and mobile divide to record their blood glucose levels.
  Arms: Arm 1; Arm 4; Arm 5; Arm 8
Behavioral: Diabetes Education Class — The diabetes education class will be administered by a certified diabetes educator.

SUMMARY:
Brief Summary:

The FREEDOM study aims to develop a scalable intervention to improve type 2 diabetes mellitus control in low-income Black adults in the Deep South. The intervention targets social determinants of health (SDoH) such as reduced healthcare access, poverty, transportation barriers, and food insecurity.

DETAILED DESCRIPTION:
Detailed Description:

1. FREEDOM Study (Type 2 Diabetes Mellitus):

   The FREEDOM study is a 12-month clinical trial enrolling 304 Black adults with Type 2 Diabetes Mellitus across three healthcare systems in Alabama and Mississippi. Participants are randomly assigned to one of eight combinations of three intervention components:
   * Digital Health Coaching: Participants receive one-on-one phone-based coaching for optimized diabetes management.
   * Food Box Delivery: Food boxes are delivered every two weeks to participants' homes,
   * Remote Patient Monitoring (RPM): Participants receive essential supplies, including glucometers, for remote blood glucose measurement. Data is monitored remotely for timely interventions.

   The study involves three in-person visits at baseline, month 6, and month 12, as well as two telephone study check-ins at month 3 and 9. Survey packets are administered at each time point.
2. FREEDOM-HIV Study (Type 2 Diabetes Mellitus and HIV Cohort):

Additionally, a cohort within the study, known as the FREEDOM-HIV study, will enroll additional 80 adults who have both Type 2 Diabetes Mellitus and HIV. This cohort will be observed over a 6-month period and will also consist of the same three intervention components.

ELIGIBILITY:
Inclusion criteria:

1. Self-identified as Black/African American
2. ICD diagnosis of T2DM
3. ≥18 years of age
4. Ongoing insulin treatment
5. HbA1c ≥8% within 6 weeks of study screening
6. has the ability to converse in and read English
7. must provide written informed consent prior to enrollment

Exclusion criteria:

1. Current enrollment in any diabetes-related interventional study
2. Cognitive impairment
3. End-stage kidney disease (CKD-5)
4. Pregnant or plans to become pregnant within 12 months
5. Currently enrolled in a structured lifestyle change program
6. Enrolled in remote patient monitoring or health coaching within 60 days of the study or intervention

HIV Cohort Criteria

Inclusion Criteria

1. ≥ 18 years of age
2. ICD diagnosis of T2DM
3. HbA1c ≥ 7%
4. Confirmed HIV+ diagnosis
5. Prescribed HIV ART therapy as part of care

Exclusion Criteria

1. Current enrollment in any diabetes-related interventional study or structured lifestyle change program
2. Enrolled in RPM or health coaching (except for coaching on smoking cessation) within 60 days of the intervention
3. Cognitive impairment
4. End-stage kidney disease (CKD-5)
5. Pregnant or plans to become pregnant within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
FREEDOM Study: Change in HbA1c level between baseline and 12 month | 12 months
  The primary outcome of the study is to track change in the HbA1c between baseline and 12 months (endpoint of the study). The HbA1C will be tested at baseline, 6 and 12 months.
Primary Outcome for the HIV Cohort: Change in HbA1c level between baseline and 6 months | 6 months
  The primary outcome of the study is to track change in the HbA1c between baseline and 6 months (endpoint of the study). The HbA1C will be tested at baseline and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Hospital and UMMC Cardiology Clinics, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Zein A, Garla V, Hall ME, Nawshin T, Hays D, John T, Delaney E, Wallace E, Hearld L, Cherrington AL, Mehta T. Rationale and design of the FREEDOM study: A hybrid type 1 optimization-implementation trial to improve type 2 diabetes management in primary care. Contemp Clin Trials. 2026 Feb;161:108173. doi: 10.1016/j.cct.2025.108173. Epub 2025 Dec 5. PMID 41354173